CLINICAL TRIAL: NCT02473523
Title: Feasibility of Implementing Yoga Intervention for Adolescents at St. Jude Children's Research Hospital
Brief Title: Yoga to Alleviate Fatigue, Anxiety and Pain in Adolescents During Treatment for Lymphoma or Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator left the institution.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: YOGAOT; NCI-2015-00975 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-06-03; First posted 2015-06-16 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Leukemia; Hodgkin Lymphoma; Lymphoma, Non-Hodgkin's
Keywords: Fatigue; Pain Alleviation; Emotional Wellbeing; Physical Wellbeing; Yoga
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Fatigue | interventions — Surveys and Questionnaires; 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participants (Experimental): Leukemia, Hodgkin Lymphoma and non-Hodgkin's Lymphoma patients who meet eligibility requirements and consent to participate in the study.
  Interventions: Yoga Therapy, PedsQL Multidimensional Fatigue Scale, PedsQL Cancer Module, Verbal Numeric Pain Scale. Biodex System 3 Dynamometer, Jamar Hydraulic Hand Dynamometer, Sit and Reach Test, and Test of Motor Proficiency.
  Interventions: Other: PedsQL Cancer Module; Other: PedsQL Multidimensional Fatigue Scale; Device: Biodex System 3 Dynamometer; Device: Jamar Hydraulic Hand Dynamometer; Other: Sit and Reach Test; Other: Test of Motor Proficiency; Other: Verbal Numeric Pain Scale; Other: :Yoga Therapy

INTERVENTIONS:
Other: PedsQL Cancer Module — The PedsQL cancer module acute version is a 27 item assessment that includes eight scales including pain (2 items), nausea (5 items), anxiety related to procedures (3 items), anxiety related to treatment (3 items), worry (3items), cognitive problems (5 items), perceived physical appearance and communication (3 items). This assessment will take approximately 15-30 minutes to complete.
  Other Names: Questionnaire
Other: PedsQL Multidimensional Fatigue Scale — The Multidimensional Fatigue Scale is an 18 item questionnaire encompassing 3 subscales including general fatigue (6 items), sleep and rest fatigue (6 items) and cognitive fatigue (6 items). This assessment will take approximately 10-20 minutes to complete.
  Other Names: Questionnaire
Device: Biodex System 3 Dynamometer — The "Biodex System 3 Dynamometer" will be used to measure isometric quadriceps muscle contractions. Participants will be stabilized in the chair with abdominal and shoulder straps. The isometric tests for knee extension will be done on both dominant and non-dominant leg. The tests consist of 3 maximal muscle contractions each lasting five seconds separated by 40 second rest intervals. This assessment will take approximately 10 minutes to complete.
  Other Names: Quadriceps Strength Measurement
Device: Jamar Hydraulic Hand Dynamometer — A calibrated "Jamar" hydraulic hand dynamometer will be used to measure grip strength. The participant will be seated in a chair with elbow flexion to 90 degrees against torso and the forearm in neutral. The participant will grasp the device and the handle will be adjusted so that digits are able to comfortably grasp the device. The maximum score after 2 trials will be recorded as grip strength for both right and left hand. This assessment will take no more than 5 minutes to complete.
  Other Names: Grip Strength Measurement
Other: Sit and Reach Test — Hamstring flexibility will be assessed by the Sit and Reach Test. The sit and reach is a test to measure hip, hamstring and lower back flexibility. To measure flexibility participants will perform the YMCA sit and reach test. Participants will sit down without shoes or socks with the soles of their feet against the vertical platform of the sit-and-reach box located at the 26 cm (a little over 10 inches) mark. Participants keep their legs straight and their hands overlapped, while reaching for a less than maximum distance twice as a warm-up. This test will take no more than 5 minutes to complete.
  Other Names: Hamstring Flexibility Measurement
Other: Test of Motor Proficiency — The Bruininks-Oseretsky Test of Motor Proficiency is a 9 item standardized assessment that includes standing with feet on a line with eyes open and closed, standing on a line with one foot with eyes open and closed, standing on a balance beam on one leg with eyes open and closed and standing heel to toe on a balance beam. These tests will be administered no more than two times with a maximum score of 10 seconds. Two additional subtests include walking forward on a line and walking heel to toe on a line for a maximum of 6 steps for both tasks. Total time to complete this test is approximately 10-20 minutes.
  Other Names: Bruininks-Oseretsky Test of Motor Proficiency; Balance Measurement
Other: Verbal Numeric Pain Scale — The verbal numeric pain scale will be administered before and after each yoga session. The principal investigator (PI) will ask the participant about his/her pain on a scale of 0-10 and the PI will record the number. This will take less than 10 seconds.
  Other Names: Pain Measurement
Other: :Yoga Therapy — Those who consent will participate in 60-minute yoga sessions 2-3 times per week for 4-6 weeks. Only specified yoga poses will be implemented during the classes. Additional detail is included in the Description sections of this registration. The principal investigator is a Certified Yoga Therapist (CYT) and is a registered yoga teacher with 500 hours of training (RYT 500).
  Other Names: Yoga Intervention; Yoga

SUMMARY:
Researchers at St. Jude Children's Research Hospital want to investigate the feasibility of a yoga intervention for adolescents receiving treatment for lymphoma or leukemia. Adolescents who participate in the program may experience improved physical and psychosocial measures. Improvements in these areas may increase participation in meaningful activity and improve quality of life.

Adolescents diagnosed with cancer may experience more fatigue, anxiety and pain during treatment. Yoga is considered a complementary alternative medicine (CAM) that has been implemented into some pediatric oncology rehabilitation programs and has been shown to be beneficial in both inpatient and outpatient settings. It may decrease anxiety and increase quality of life and hamstring flexibility in teens.

PRIMARY OBJECTIVE:

* To determine the feasibility of yoga intervention for adolescents during lymphoma and leukemia treatment.

OTHER PRE-SPECIFIED OBJECTIVE:

* To obtain pilot data regarding efficacy of yoga on pain, quality of life, fatigue and physical performance.

DETAILED DESCRIPTION:
Those who consent to participate will participate in 60-minute yoga sessions 2-3 times per week for 4-6 weeks. Only specified yoga poses will be implemented during the classes.

The study will be done in three parts: initial evaluation, yoga therapy, and follow-up evaluations.

INITIAL EVALUATION: Participants will complete the PedsQL Cancer Module questionnaire and the PedsQL Multidimensional Fatigue Scale questionnaire. Physical performance including quadriceps strength, grip strength, hamstring flexibility, and balance, will be assessed.

YOGA THERAPY: The principal investigator (PI) is a certified yoga therapist (CYT) and is a registered yoga teacher with 500 hours of training (RYT 500). Participants will take part in a 60-minute yoga session conducted by the PI 2-3 times a week for 4-6 weeks, during which time they must complete 8-12 yoga sessions. The yoga intervention includes these parts: warm-up, strengthening, increasing hamstring flexibility, balance and relaxation. Yoga poses will be used for each yoga session from a predetermined roster depending on individual adolescent abilities. This will allow for a tailored but standardized yoga intervention. Modifications including chairs, straps and blocks will be allowed to promote appropriate form and use of these props will be recorded. Immediately before and after each yoga session, the therapist will record pain with the verbal numeric pain scale.

FOLLOW-UP EVALUATIONS: After completion of the 4-6 weeks of yoga therapy, participants will complete all assessments and physical performance measures that were done in the initial evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient being treated at St. Jude Children's Research Hospital
* Diagnosis of lymphoma or leukemia as documented in medical record
* Physician approval to participate in intervention
* Ages 13-17 years
* Ability to come to standing from seated position without assistance
* Parent or legal guardian consent
* Adolescent gives assent
* English speaking

Exclusion Criteria:

* Participant not planning on remaining at St Jude for at least 4 weeks
* Cognitive impairment that prevents participant from answering questions in standardized assessments

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Doria Braman, MSOT, OTR/L, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants were enrolled between February and April 2016.
Groups:
- Participants: Leukemia, Hodgkin Lymphoma and non-Hodgkin's Lymphoma patients who meet eligibility requirements and consent to participate in the study.
  Participants were to undergo the following interventions: Yoga Therapy, PedsQL Multidimensional Fatigue Scale, PedsQL Cancer Module, Verbal Numeric Pain Scale. Biodex System 3 Dynamometer, Jamar Hydraulic Hand Dynamometer, Sit and Reach Test, and Test of Motor Proficiency.
Period: Overall Study
Arm/Group | Participants
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 0
Age, Continuous
Gender

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients Who Are Willing to Participate
Description: The rate of participants who are willing to participate on this protocol to the total number of participants approached. It is anticipated that 50% approached patients will agree to participate on the study. Twenty five patients will be approached and asked to participate in the study. If more than 6 patients out of 25 approached patients refuse to participate in the study, the study will be closed, and it will be concluded that the trial is not feasible.
Time Frame: Day 0
Arm/Group | Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Rate of Patients Who Complete the Study
Description: The rate of enrolled and consented patients who complete the 60-minute yoga sessions offered over a 4-6 week period to the total number of participants on the study. It is hypothesized that 60% of those participants will complete the intervention. Thus, if more than 5 patients can not complete the intervention, then it will be concluded that the trial is not feasible.
Time Frame: At end of 4-6 weeks
Arm/Group | Participants
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Mean Change in PedsQL Cancer Module Score
Description: Mean ± standard error will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Median Change in PedsQL Cancer Module Score
Description: Median (range) will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Mean Change in PedsQL Multidimensional Fatigue Scale
Description: Mean ± standard error will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Median Change in PedsQL Multidimensional Fatigue Scale
Description: Median (range) will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Mean Change in Quadriceps Strength
Description: The "Biodex System 3 Dynamometer" will be utilized to measure isometric quadriceps muscle contractions. Mean ± standard error will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Median Change in Quadriceps Strength
Description: The "Biodex System 3 Dynamometer" will be utilized to measure isometric quadriceps muscle contractions. Median (range) will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Mean Change in Grip Strength
Description: A calibrated "Jamar" hydraulic hand dynamometer will be used to measure grip strength. Mean ± standard error will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Median Change in Grip Strength
Description: A calibrated "Jamar" hydraulic hand dynamometer will be used to measure grip strength. Median (range) will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Mean Change in Hamstring Flexibility
Description: Hamstring flexibility will be assessed by the Sit and Reach Test. Mean ± standard error will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Median Change in Hamstring Flexibility
Description: Hamstring flexibility will be assessed by the Sit and Reach Test. Median (range) will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Mean Change in Balance
Description: Mean ± standard error on the Bruininks-Oseretsky Test of Motor Proficiency will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Median Change in Balance
Description: Median (range) on the Bruininks-Oseretsky Test of Motor Proficiency will be provided.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Mean Change in Verbal Numeric Pain Scale
Description: Summary statistics of mean ± standard error will be provided. Longitudinal change for the numeric pain scale across the yoga session will be reported.
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Median Change in Verbal Numeric Pain Scale
Description: as for outcome 15
Time Frame: Baseline at initial evaluation to follow-up evaluation (up to 6 weeks later)
Arm/Group | Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were to be recorded from the on-study date until the participant was taken off study, a maximum of 6 weeks.
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated because the principal investigator left the institution. One participant completed only 8 of 16 sessions and was not evaluable for study objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes